CLINICAL TRIAL: NCT04224896
Title: Narrow-Band Imaging (NBI) Versus Lugol Chromoendoscopy in the Detection of Oesophagus Squamous Cell Carcinoma in High Risk Population: a Randomised Controlled Multicentre Trial
Brief Title: Narrow-Band Imaging (NBI) Versus Lugol Chromoendoscopy in the Detection of Oesophagus Squamous Cell Carcinoma in High Risk Population
Status: Completed | Type: Observational
Sponsor: Hôpital Edouard Herriot (Other)
Responsible Party: Principal Investigator, Jean Christophe Saurin, Professor, Hôpital Edouard Herriot
Other Study IDs: SFED
Record Dates: First submitted 2020-01-08; First posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: FRENCH STUDY
MeSH Terms: interventions — Gastroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NBI PATIENT
  Interventions: Diagnostic Test: UPPER ENDOSCOPY
- LUGOL PATIENT
  Interventions: Diagnostic Test: UPPER ENDOSCOPY

INTERVENTIONS:
Diagnostic Test: UPPER ENDOSCOPY — UPPER ENDOSCOPY

SUMMARY:
Narrow-Band Imaging (NBI) is as sensitive as Lugol chromoendoscopy to detect oesophageal squamous cell carcinoma (SCC) and appears more specific than Lugol chromoendoscopy in expert centres but its specificity in current practice is not known. This study aimed to prove the superiority of NBI specificity over Lugol chromoendoscopy to detect oesophageal SCC and high-grade dysplasia (HGD) in current practice (including tertiary care centres, local hospitals and private clinics).

ELIGIBILITY:
Inclusion Criteria:

* Patients had a history or current SCC

Exclusion Criteria:

* NONE

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: HIGH RISK OF OESOPHAGEAL SQUAMOUS CELL CARCINOMA
Sampling Method: Non-Probability Sample
Enrollment: 335 (Actual)
Dates: Start 2011-03-01 (Actual); Primary Completion 2011-03-01 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
SPECIFICITY OF THE TWO DIAGNOSTIC STRATEGIES | 4 years

REFERENCES:
- [Derived] Gruner M, Denis A, Masliah C, Amil M, Metivier-Cesbron E, Luet D, Kaasis M, Coron E, Le Rhun M, Lecleire S, Antonietti M, Legoux JL, Lefrou L, Renkes P, Tarreirias AL, Balian P, Rey P, Prost B, Cellier C, Rahmi G, Samaha E, Fratte S, Guerrier B, Landel V, Touzet S, Ponchon T, Pioche M. Narrow-band imaging versus Lugol chromoendoscopy for esophageal squamous cell cancer screening in normal endoscopic practice: randomized controlled trial. Endoscopy. 2021 Jul;53(7):674-682. doi: 10.1055/a-1224-6822. Epub 2020 Oct 1. PMID 32698233